CLINICAL TRIAL: NCT01415674
Title: Multi-centric Randomized Phase II Study of Pre-operative Afatinib (BIBW2992) Aiming at Identifying Predictive and Pharmacodynamic Biomarkers of Biological Activity and Efficacy in Untreated Non-metastatic Head and Neck Squamous Cell Carcinoma Patients
Brief Title: Research of Biomarkers of Activity and Efficacy of BIBW2992 in Untreated Non-metastatic HNSCC Patients
Acronym: PREDICTOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEP11/1010
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck
Keywords: Squamous cell carcinoma of the head and neck; pre operative treatment; Afatinib; BIBW2992; Biological markers
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Afatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Afatinib 40mg per os daily (Experimental): Patients randomized to the arm A will take a single oral dose of Afatinib from Day 1, for 14 to 28 days, depending on the date of surgery. The number of dosing days will be chosen so that patients are off treatment for a maximum of 7 days before surgery.
  Interventions: Drug: Afatinib
- Arm B : No pre operative treatment (No Intervention)

INTERVENTIONS:
Drug: Afatinib — Afatinib 40mg per os daily for 14 to 28 days, depending on the date of the surgery
  Other Names: BIBW2992
  Arms: Arm A: Afatinib 40mg per os daily

SUMMARY:
The purpose of this study is to identify predictive and pharmacodynamic biomarkers of activity and efficacy of pre-operative Afatinib (BIBW2992) in untreated non-metastatic head and neck squamous cell carcinoma patients

DETAILED DESCRIPTION:
More than 500,000 new patients with squamous cell carcinomas of the head and neck (SCCHN) are diagnosed each year around the world. Patients who relapse after primary therapy for locoregional disease and those who present with distant metastases have limited prognosis.

Drug therapy for cancer control and the palliation of patients with recurrent or metastatic SCCHN is currently suboptimal. In contemporary trials the most active cytotoxic drug combinations have response rates in the range of 30%, and are associated with frequent and severe toxicities and treatment-related mortality.

Molecular targeting has been demonstrated in oncology as a relevant strategy in cancer therapeutics. In March 2006, the FDA announced the approval of a chimeric monoclonal antibody against the epidermal growth factor receptor (EGFR), cetuximab, for use in combination with radiation therapy in patients with locally advanced SCCHN. Furthermore, the addition of cetuximab to cisplatin and 5FU as first-line therapy in patients with recurrent or metastatic SCCHN has significantly improved overall survival when compared to cisplatin and 5FU alone. Phase II data of cetuximab given as monotherapy in recurrent or metastatic SCCHN patients who have progressed on platinum-based therapy have demonstrated an overall response rate of 13% and a median survival of about 6 months. Small molecules tyrosine kinase inhibitors of EGFR, such as gefitinib and erlotinib, seem to be slightly less effective than cetuximab. Based on these results, FDA has also approved cetuximab monotherapy use for this indication in recurrent or metastatic SCCHN.

However, despite high expression of EGFR in SCCHN, EGFR inhibitor monotherapy has only had modest activity. Potential mechanisms of resistance to EGFR-targeted therapies involve EGFR and K-Ras mutations, epithelial-mesenchymal transition, and activation of alternative and downstream pathways. Strategies to optimize EGFR-targeted therapy in head and neck cancer involve the selection for patients most likely to benefit and the use of therapies to target the network of pathways involved in tumor growth, invasion, angiogenesis, and metastasis.

Afatinib is an irreversible dual inhibitor of EGFR and HER2 tyrosine kinase. Preclinical data suggest that Afatinib might have a larger spectrum antitumor activity than EGFR tyrosine kinase inhibitors. In vivo and in vitro studies indeed showed that Afatinib displays antitumor activity in erlotinib/gefitinib-resistant lung models. Afatinib compared favourably to cetuximab in platinum-resistant metastatic SCCHN. In addition, Afatinib has shown promising antitumor activity in HER2-overexpressing metastatic breast cancer after trastuzumab failure and in metastatic adenocarcinomas of the lung harbouring EGFR activating mutations.

To date, predictive and pharmacodynamic biomarkers studies have mostly been performed in pre-treated metastatic patients. Erlotinib has been the most studied EGFR-targeted agent in terms of biomarkers identification in SCCHN. In the metastatic setting, sequential biopsies allowed correlating potential predictive and pharmacodynamic biomarkers with the outcome of patients treated with erlotinib. The decrease of p-EGFR in tumor tissue was associated with increased time-to-progression (TTP) and overall survival (OS) in one study. In another study, elevated pre-treatment levels of p27 and p-STAT3 in tumor tissue predicted for prolonged TTP and OS, while a decrease in p-EGFR, p-NFkB and p27 correlated with increased TTP, OS or both. However, the lack of control arm precluded to draw any definitive conclusion. One study evaluated erlotinib in the neoadjuvant setting in untreated patients with operable SCCHN. Baseline p21 expression in tumor tissue correlated with clinical response to treatment. But again, the absence of control arm in this later study precluded drawing definitive conclusions regarding the potential predictive and pharmacodynamic value of the biomarkers under evaluation.

The main characteristics of our study are:

1. the pre-operative setting in untreated patients with the advantage of having untreated patients for whom it is easy to get pre- and post-treatment tumor specimen, during initial panendoscopy and surgery, respectively
2. the randomization versus no treatment which is the only way to be able to draw robust conclusions regarding the potential predictive and pharmacodynamic value of the biomarkers under evaluation. Single-arm phase II trials can only identify prognostic markers of activity, but not predictive biomarkers of activity.

Importantly, surgery will not be delayed in any case by the study. However, it is required that planning of surgery will enable patients to receive between 21 and 28 days of treatment to participate into the study given the planned date of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, larynx or hypopharynx, previously untreated, amenable to curative treatment with surgery. Patients with a diagnosis of SCCHN of occult primary may be enrolled only with the agreement of the lead investigator upon review of the relevant clinical records
* T2-4N0-2 tumors (except T2N0 endolaryngeal tumors)
* Absence of metastases determined by PET CT scan
* Planned date of surgery allowing the patient to receive between 21 and 28 days of treatment
* ECOG performance status ≤ 2
* Adequate bone marrow function (absolute neutrophil count > 1,000 cells/mm³, platelets > 75,000 cells/mm³)
* Adequate liver function (total bilirubin ≤ 1.5 x UNL [upper normal limit], AST or ALT ≤ 3 x UNL)
* Adequate renal function (serum creatinine ≤ 1.5 x UNL)
* Adequate cardiac function (a normal left ventricular ejection fraction [LVEF] of ≥ 50% as measured by MUGA scan or echocardiogram within 4 weeks prior to start of study treatment)
* Potentially reproductive patients must agree to use an effective contraceptive method while on treatment
* Women of childbearing potential must have a negative serum beta-HCG pregnancy test within 7 days prior of enrollment and/or urine pregnancy 48 hours prior to the administration of the first study treatment
* Patients must be able to swallow tablets
* Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
* Patients must be affiliated to a Social Security System
* Patient information and written informed consent form signed

Exclusion Criteria:

* Primary site of head and neck carcinoma in nasopharynx, or skin
* T1N0 tumors and T2N0 endolaryngeal tumors
* Patients not candidate for primary curative surgery
* Planning of surgery not allowing the patient to receive 21 to 28 days of treatment
* Patients receiving other anti-cancer medication such as chemotherapy, immunotherapy, biologic therapy or hormonal therapy (other than leuprolide or other GnRH agonists) within 30 days prior to the first dose of study drug and while on study treatment.
* Patients receiving other anti-cancer non-drug therapies: radiation, or tumor embolization within 4 weeks prior to the first dose of study drug and while on study treatment.
* Patient being treated with anti-vitamin K (AVK). Low molecular weight heparin (LMWH) is allowed.
* Patient with uncontrolled infection
* Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study, including uncontrolled diabetes,
* Clinically relevant cardiovascular abnormalities, as judged by the investigator, such as, but not limited to, uncontrolled hypertension, congestive heart failure NYHA classification > III, unstable angina, myocardial infarction within six months prior to randomisation, or poorly controlled arrhythmia, chronic liver or renal disease, severely impaired lung function
* Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g. Crohn's disease, malabsorption or CTCAE grade >1 diarrhea of any etiology at randomisation
* Known pre-existing Interstitial Lung Disease (ILD)
* Patients requiring comedication with potent P-gp inhibitors (including Cyclosporin, Erythromycin, Ketoconazole, Itraconazole, Quinidine, Phenobarbital salt with Quinidine, Ritonavir, Valspodar, Verapamil) or inducers (including St John's wort, rifampicin)
* Patients with a known HIV, active hepatitis B and/or C infection
* Pregnant women, women who are likely to be pregnant or are breast-feeding
* Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Patients who received any other investigational drugs within 30 days prior to the screening visit and/or during the study
* Patients unwilling to participate in the biological investigations
* Individually deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Potential predictive biological markers of activity of Afatinib | 15 days (FDG-PET evaluation) and about 21 days (CT scan or MRI evaluation) after start of treatment
  Correlation between baseline potential biomarkers and
  1. radiological response to Afatinib
  2. FDG-PET response to Afatinib
  To identify the predictive biomarkers, the following translational researches will be carried out on initial tumor biopsy
  * IHC tumour characterization
  * High throughput protein analysis
  * Molecular analyses : FISH , Mutations by PCR , Quantitative RT-PCR

SECONDARY OUTCOMES:
Potential pharmacodynamic biological markers of activity of Afatinib | 15 days (FDG-PET evaluation) and about 21 days (CT scan or MRI evaluation) after start of treatment
  Correlation between down- or up-regulation of potential biomarkers (in pre-treatment biopsy and surgical specimen) and
  1. radiological response to Afatinib
  2. FDG-PET response to Afatinib
  To identify the pharmacodynamic biomarkers, the following translational researches will be carried out on initial tumor biopsy and surgical specimen
  * IHC tumour characterization
  * High throughput protein analysis
  * Molecular analyses : FISH , Mutations by PCR , Quantitative RT-PCR
Efficacy of Afatinib | about 21 days (CT scan or MRI evaluation) after start of treatment
  - Efficacy will be defined as the tumour reduction between the baseline and the surgery (end of treatment). The radiological response will be assessed on CT/MRI of the head and neck. Tumour size will be the sum of 2 target lesions following the measurement rules from the RECIST 1.1. Noteworthy, a lymph node can be considered a target lesion only if its smallest diameter is ≥15 mm (according to RECIST 1.1). Measurement of a lymph node consists in measuring its smallest diameter (according to RECIST 1.1).
Toxicity of Afatinib | every week until surgery.
  Toxicity will be assessed according to NCI CTC-AE v4.0 criteria
Pathological response | on the surgical specimen
  Complete pathological response is defined as the absence of invasive cancer cells on the surgical specimen in the primary tumor and in lymph nodes.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Le Tourneau, Principal Investigator — Institut Curie Paris
Locations (11):
- France (11):
  - CHU d'Angers, Angers
  - Institut de cancérologie de l'Ouest - Site Paul Papin, Angers
  - Centre François Baclesse, Caen
  - Centre Léon Bérard, Lyon
  - Chu de Nantes, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut de cancérologie de l'Ouest - Site René Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif